CLINICAL TRIAL: NCT02145299
Title: A Prospective, Multicenter, Open Label Randomized Study to Evaluate the Safety, Performance and Intraluminal Crossing of the TruePath™ CTO Device Versus The Crosser System in Patients With Symptomatic Femoro-popliteal Chronic Total Occlusion (CTO)
Brief Title: The Lumen Study: Comparing Devices for Patients With Symptomatic Femoro-popliteal Chronic Total Occlusion (CTO)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was stopped due to insufficient numbers of subjects to meet study design objectives.
Sponsor: Yale University (Other)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HIC140101333
Record Dates: First submitted 2014-05-19; First posted 2014-05-22 (Estimated); Results first posted 2016-11-04 (Estimated); Last update posted 2016-11-04 (Estimated); Status verified 2016-09

CONDITIONS: Symptomatic Femoro-popliteal Chronic Total Occlusion

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- TruePath CTO Device (Experimental): The TruePath™ CTO Device (Boston Scientific Corporation, Natick, MA) is a new solution for intraluminal treatment of chronic total occlusions (CTO). It is the longest available crossing device (165 cm), and has a diamond-coated distal tip that can rotate at 13,000 rpm. Its profile is similar to a 0.018" guidewire, and includes a shapeable distal tip allowing 1:1 torque response. In addition, it provides audio and visual navigation during CTO crossing.
  Interventions: Device: TruePath CTO Device
- CROSSER CTO Device (Active Comparator): The CrosserTM CTO Recanalization Catheter ("Crosser system") (Bard Peripheral Vascular Inc. Tempe, AZ, USA), which serves as a control in this investigation, gained U.S. FDA approval for peripheral indications in 2011. The device is similar in both design and indications to the TruePath device, with the exception that the Crosser system uses vibrational angioplasty to achieve CTO crossing.
  Interventions: Device: CROSSER CTO Device

INTERVENTIONS:
Device: TruePath CTO Device — The TruePath CTO Device is composed of a 0.018" guidewire and a motor housing with a connector cable along with a sterile, disposable battery-powered Control Unit for manipulation of the device during operation. The TruePath CTO Device is indicated to facilitate the intra-luminal placement of conventional guidewires beyond peripheral artery chronic total occlusions.
  Arms: TruePath CTO Device
Device: CROSSER CTO Device
  Arms: CROSSER CTO Device

SUMMARY:
This is a prospective, multicenter, randomized, single-blind study enrolling up to 75 subjects at up to 5 sites in the US. Eligible subjects with symptomatic femoro-popliteal CTO will be randomized 2:1 to treatment with the TruePath™ CTO Device (Intervention) or the CROSSER™ CTO device (Control). All patients will receive standard anticoagulation per hospital protocol and antiplatelet therapy with aspirin and clopidogrel.

DETAILED DESCRIPTION:
The primary objective of the study is to compare the technical success and in-hospital safety of TruePath device with that of the CROSSER device in patients with symptomatic femoro-popliteal CTO. Subjects will be followed clinically while in the hospital and at 1 month following the index procedure. All subjects will undergo procedural intravascular ultrasound (IVUS) imaging. The study population will consist of up to 75 patients with symptomatic femoro-popliteal CTO and indications for revascularization. Subjects must have a previously documented conventional percutaneous procedure or a concurrent failed attempt to cross the CTO using conventional guidewire techniques. All subjects must meet all inclusion and no exclusion criteria and sign an Informed Consent Form approved by the local Institutional Review Board (IRB) prior to enrollment and randomization.

ELIGIBILITY:
Inclusion Criteria:

* Clinical Inclusion Criteria
* Male or non-pregnant female ≥18 years of age;
* Rutherford Clinical Category 2-5
* Patients is willing to provide informed consent and comply with the required follow-up visits, testing schedule, and medication regimen
* Angiographic Lesion Inclusion Criteria
* Length ≤35 cm
* The lesion is a single lesion or composite of multiple lesions within the 35 cm segment
* 100% stenosis by visual estimate
* Previously documented conventional percutaneous procedure or a concurrent failed attempt to cross the CTO using conventional guidewire techniques
* Ability to visualize target artery distal to the lesion (via collateral circulation)
* Target lesion located in the superficial femoral/proximal popliteal arteries, with lesion location starting ≥1cm below the common femoral bifurcation
* De novo lesion or restenotic lesion >30 days from any prior endovascular intervention
* Target vessel diameter ≥4 and ≤7 mm and able to be treated with PTA and or a stent
* A patent inflow artery free from significant lesions (≥50% stenosis) as confirmed by angiography. Treatment of the target lesion may be performed after successful treatment of existing inflow artery lesions at the time of the index procedure. [NOTE: Successful inflow artery treatment is defined as attainment of residual diameter stenosis ≤50% without death or major vascular complication.]
* At least one patent outflow artery free from significant lesion (≥50% stenosis) as confirmed by angiography (treatment of outflow disease is permitted)

Exclusion Criteria:

* Pregnant or nursing subjects and those who plan pregnancy in the period up to 3 months following index procedure. Female subjects of child-bearing potential must have a negative pregnancy test done prior to the index procedure.
* Rutherford Class 0, 1 or 6
* History of hemorrhagic stroke within 3 months
* Renal failure or chronic kidney disease with MDRD GFR ≤ 30 ml/min per 1.73m2 (or serum creatinine ≥2.5 mg/L within 30 days of index procedure or treated with dialysis)
* Previous or planned surgical or interventional procedure to the target limb within 2 weeks before (aside from conventional percutaneous procedure during the current hospitalization) or within 30 days after the index procedure
* Prior vascular surgery of the index limb, with the exception of common femoral patch angioplasty remote from the target lesion
* Planned use of adjunctive primary treatment modalities (e.g., laser, atherectomy, cryoplasty, scoring/cutting balloon, or other)
* Inability to take required study medications or an allergy to contrast that cannot be controlled with medication
* Life expectancy of <1 years
* Patient is currently participating in an investigational drug or device study or previously enrolled in this study Subject enrollment and treatment

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2014-05; Primary Completion 2015-03 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Mena, MD, Principal Investigator — Yale University; Alexandra Lansky, MD, Principal Investigator — Yale University
Locations (1):
- Yale Cardiovascular Research Group, New Haven, Connecticut, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- CROSSER CTO Device: The CrosserTM CTO Recanalization Catheter ("Crosser system") (Bard Peripheral Vascular Inc. Tempe, AZ, USA), which serves as a control in this investigation, gained U.S. FDA approval for peripheral indications in 2011. The device is similar in both design and indications to the TruePath device, with the exception that the Crosser system uses vibrational angioplasty to achieve CTO crossing.
  CROSSER CTO Device
Period: Overall Study
Arm/Group | TruePath CTO Device | CROSSER CTO Device
Started | 6 | 2
Completed | 6 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Only 8 subjects were recruited and enrolled overall- study was terminated.
Groups:
- Total: Total of all reporting groups
Arm/Group | TruePath CTO Device | CROSSER CTO Device | Total
Number analyzed (Participants) | 6 | 2 | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.0 (7.1) | 64.0 (11.0) | 67.8 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 5 | 2 | 7

OUTCOME MEASURES:

1. Primary Outcome: Technical Success
Description: Technical success, defined as the ability to facilitate complete intraluminal crossing of a CTO into the true distal lumen with a TruePath or a CROSSER device and/or any subsequent conventional guidewire, as confirmed by IVUS imaging
Time Frame: Day of operation
Measure: Number; unit: percentage of participants
Arm/Group | TruePath CTO Device | CROSSER CTO Device
Number analyzed (Participants) | 6 | 2
percentage of participants | 50 | 0

2. Primary Outcome: In-hospital Safety
Description: In-hospital safety, defined as a composite of all-cause death, index limb amputation above the ankle, and target lesion revascularization (TLR)
Time Frame: Operation through 30 day follow up
Measure: Number; unit: percentage of participants
Arm/Group | TruePath CTO Device | CROSSER CTO Device
Number analyzed (Participants) | 6 | 2
percentage of participants | 0 | 0

3. Secondary Outcome: Procedural Success
Description: Procedural success, defined as technical success and (1) residual stenosis <50% in the treated segment (2) and improved distal flow by angiography following the procedure
Time Frame: Day of operation
Population: Due to early study termination for reason unrelated to safety, rather enrollment challenges, part the Procedural Success definition required % residual stenosis which was going to be a Core Laboratory assessment to eliminate bias and maintain consistency in the analysis. With only 8 subjects enrolled, laboratory analysis was not undertaken.
Arm/Group | TruePath CTO Device | CROSSER CTO Device
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Clinical Success
Description: Clinical Success defined as procedure success in the absence of in-hospital all-cause death, index limb amputation above the ankle, and TLR.
Time Frame: Day of operation
Population: These data were not fully captured and summarized as the study was terminated.
Arm/Group | TruePath CTO Device | CROSSER CTO Device
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Symptomatic Improvement
Description: Symptomatic improvement, as assessed by change in Rutherford Class from baseline to 30 days
Time Frame: Baseline, and 30 days post operation
Measure: Number; unit: percentage of participants
Arm/Group | TruePath CTO Device | CROSSER CTO Device
Number analyzed (Participants) | 6 | 2
percentage of participants | 50 | 50

6. Secondary Outcome: Walking Capacity
Description: Change in walking capacity from baseline to 30 days, measured by the Walking Impairment Questionnaire. The questionaire is a subjective measure of patient-perceived walking performance developed for individuals with peripheral arterial disease. Used to evaluate the "change in walking capacity" study endpoint.
Time Frame: Baseline and 30 days post operation
Population: These data were not fully captured and summarized as the study was terminated.
Arm/Group | TruePath CTO Device | CROSSER CTO Device
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Index Limb Amputation
Description: Need for limb amputation
Time Frame: Day of Operation through 30 days post operation
Measure: Number; unit: participants
Arm/Group | TruePath CTO Device | CROSSER CTO Device
Number analyzed (Participants) | 6 | 2
participants | 0 | 0

8. Secondary Outcome: Target Lesion Revascularization
Description: Describes the percentage of patients that had stented lesions that had to be re-treated due to clinically-driven restenosis.
Time Frame: 30 days post operation
Measure: Number; unit: percentage of participants
Arm/Group | TruePath CTO Device | CROSSER CTO Device
Number analyzed (Participants) | 6 | 2
percentage of participants | 0 | 0

9. Secondary Outcome: Ankle-brachial Index (ABI)
Description: The ratio of systolic blood pressure at the ankle to systolic blood pressure in the arm
Time Frame: baseline to 30 days post operation
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | TruePath CTO Device | CROSSER CTO Device
Number analyzed (Participants) | 6 | 2
ratio
  Baseline | 0.63 (0.18) | 0.75 (0.19)
  30 days | 0.68 (0.24) | 0.93 (0.07)

10. Secondary Outcome: Target Vessel Revascularization
Description: A repeat revascularization procedure (percutaneous or surgical) of the index procedure target vessel. TVR is classified as clinically-driven if the repeat intervention is driven by clinical findings (ischemic symptoms).
Time Frame: 30 days post operation
Measure: Number; unit: percentage of participants
Arm/Group | TruePath CTO Device | CROSSER CTO Device
Number analyzed (Participants) | 6 | 2
percentage of participants | 16.7 | 0

11. Secondary Outcome: Angiographic Perforation Classification and Rate
Description: Evaluated in-hospital. The occurrence of any extravasation of contrast during the procedure (detected by the physician performing the procedure, or preferentially the Angiographic Core Laboratory) will be tabulated according to the standard Type 1-3 classification. Type 1 - Extraluminal crater without contrast extravasation
  * Type 2 - Perivascular blush without contrast jet extravasation
  * Type 3 - Contrast jet extravasation through frank (≥1 mm) perforation
Time Frame: Day of operation
Population: These data were not fully captured and summarized as the study was terminated.
Arm/Group | TruePath CTO Device | CROSSER CTO Device
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | TruePath CTO Device | CROSSER CTO Device
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/2
Other Adverse Events (participants affected / at risk) | 0/6 | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes